CLINICAL TRIAL: NCT04451642
Title: A Retrospective Clinical Registry of Peripheral Nerve Block: Current Practice and Complications
Brief Title: A Retrospective Clinical Registry of Peripheral Nerve Block
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria Aragón (Other)
Collaborators: Hospital Miguel Servet (Other)
Responsible Party: Sponsor
Other Study IDs: POF-LEV-2019-01
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2020-06

CONDITIONS: Nerve Block; Regional Anesthesia; Postoperative Complications
Keywords: Regional Anesthesia; Postoperative neurological complications; Ultrasound; Nerve stimulator; Brachial Plexus Block
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Peripheral nerve block Group: Every patient scheduled during 2011-2019 for the surgery needed a peripheral nerve block were enrolled.
  Interventions: Procedure: Peripheral nerve block

INTERVENTIONS:
Procedure: Peripheral nerve block — Peripheral nerve block consists of the administration of a local anaesthetic into the nerves to inhibit nerve transmission in a specific part of the body. Ultrasound or Nerve stimulator could be used to locate the peripheral nerve. A needle is placed through the anatomical references to administer local anaesthetic around the peripheral nerve. Single-shot or continuous blocks are performed preoperatively and postoperatively as current practice in the surgery theatre. Using ultrasound, in-plane or out-plane approach could be performed. Peripheral nerve block provides excellent intraoperative and postoperative analgesia decreasing the need for intravenous pain drugs. Interscalene block, supraclavicular block, safene block, femoral block, BRILMA block are different kinds of peripheral nerve block using in the anaesthestic current practice.

SUMMARY:
Locorregional anaesthesia have been increased its role in different kind of surgeries, alone or combined with general anesthesia. Due to ultrasound, peripheral nerve blocks have been increased their importance in locoregional anaesthesia. They provide excellent intraoperative and postoperative analgesia, decreasing the need for intravenous opioids which increase postoperative nausea and vomiting which may prolong hospital stay.

The primary study objective is to analyze retrospectively the use of peripheral nerve blocks in the current practice of a specialized regional anaesthesia division.

This is an observational, retrospective and unicenter study. 1346 patients scheduled for the surgery needed a peripheral nerve block were enrolled.

DETAILED DESCRIPTION:
Locorregional anaesthesia have been increased its role in different kind of surgeries, alone or combined with general anesthesia. Due to ultrasound, peripheral nerve blocks have been increased their importance in locoregional anaesthesia. They provide excellent intraoperative and postoperative analgesia, decreasing the need for intravenous opioids which increase postoperative nausea and vomiting which may prolong hospital stay.

However, peripheral nerve blocks may be associated with postoperative complications, especially neurological ones. Classically, interscalene brachial plexus block produced a 100% incidence of phrenic nerve paralysis with resultant pulmonary compromise. Little literature has published a following of complications.

The primary study objective is to analyze retrospectively the use of peripheral nerve blocks in the current practice of a specialized regional anaesthesia division. The secondary objectives are assessed the patients characteristics of our sample, local anaesthetic dose used, the peripheral nerve block operator, the nerve location technique, the surgery and the complication rate after peripheral nerve block.

This is an observational, retrospective and unicenter study. 1346 patients scheduled for the surgery needed a peripheral nerve block were enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Every patient who needs a peripheral nerve block performed by Anestesia Department.

Exclusion Criteria:

* Patient refusal of peripheral nerve block.
* Known allergy to amide local anaesthetic drugs
* Absolute contraindications to perform a peripheral nerve block as coagulopathy, active infection at the block site or severe respiratory background.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited from the current practice of the Anesthesia Department (Division of Regional Anesthesia) at the Hospital Universitario Miguel Servet (HUMS) in Zaragoza, Spain. HUMS provides health care to a population size of about 400000 inhabitants, mostly urban, and more than 200 shoulder and upper extremity surgeries are performed every year.
Sampling Method: Non-Probability Sample
Enrollment: 13816 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Peripheral nerve block | During procedure
  This primary outcome is the type of peripheral nerve block performed
Incidence and frequency of Serious Adverse Events (SAE) | From performing the peripheral nerve block to 1-year follow-up
  This primary outcome is the incidence, frequency and severity of Serious Adverse Events (SAE) as assessed by CTCAE v4.0 after peripheral nerve block.

SECONDARY OUTCOMES:
Incidence and frequency of Postoperative neurological complications (PONC) | From performing the peripheral nerve block to 1-year follow-up
  This secondary outcome is the incidence, frequency and severity of Postoperative neurological complications (PONC) as assessed by CTCAE v4.0 after peripheral nerve block.
Local anesthetic used in peripheral nerve block | During procedure
  Local anesthetic type (FDA drug) used in peripheral nerve block performance
Local anesthetic dose used in peripheral nerve block | During procedure
  Local anesthetic dose (mg) used in peripheral nerve block performance
Local anesthetic volume used in peripheral nerve block | During procedure
  Local anesthetic volume (ml) used in peripheral nerve block performance
Nerve location technique used in peripheral nerve block | During procedure
  Type of nerve location technique (ultrasound, nerve stimulator or paresthesia techinique) used in peripheral nerve block performance
Peripheral nerve block operator | During procedure
  Anesthesiologist operator of peripheral nerve block (attending or trainee).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Oliver Forniés, MD, Principal Investigator — Hospital Miguel Servet
Locations (1):
- Hospital Universitario Miguel Servet, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD will be available on file in storage and on the Internet (URL undecided yet) after finishing the data collection for 25 years at the participating site.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting in July 2021 for 25 years. DOI: 10.1007/s00540-021-02989-7
Access Criteria: * To contact to Study Principal Investigator.
  * To provide to Study Principal Investigator a request to explain the reason to access to IPD study.
URL: https://click.endnote.com/viewer?doi=10.1007%2Fs00540-021-02989-7&token=WzMwOTc0MjEsIjEwLjEwMDcvczAwNTQwLTAyMS0wMjk4OS03Il0.Mx20LMo0vR9ZI0CnH8cJ4g7lBD8

REFERENCES:
- [Background] Toma O, Persoons B, Pogatzki-Zahn E, Van de Velde M, Joshi GP; PROSPECT Working Group collaborators. PROSPECT guideline for rotator cuff repair surgery: systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2019 Oct;74(10):1320-1331. doi: 10.1111/anae.14796. Epub 2019 Aug 7. PMID 31392721
- [Background] Singh A, Kelly C, O'Brien T, Wilson J, Warner JJ. Ultrasound-guided interscalene block anesthesia for shoulder arthroscopy: a prospective study of 1319 patients. J Bone Joint Surg Am. 2012 Nov 21;94(22):2040-6. doi: 10.2106/JBJS.K.01418. PMID 23172321
- [Background] Auroy Y, Benhamou D, Bargues L, Ecoffey C, Falissard B, Mercier FJ, Bouaziz H, Samii K. Major complications of regional anesthesia in France: The SOS Regional Anesthesia Hotline Service. Anesthesiology. 2002 Nov;97(5):1274-80. doi: 10.1097/00000542-200211000-00034. PMID 12411815
- [Background] Bomberg H, Wetjen L, Wagenpfeil S, Schope J, Kessler P, Wulf H, Wiesmann T, Standl T, Gottschalk A, Doffert J, Hering W, Birnbaum J, Kutter B, Winckelmann J, Liebl-Biereige S, Meissner W, Vicent O, Koch T, Burkle H, Sessler DI, Volk T. Risks and Benefits of Ultrasound, Nerve Stimulation, and Their Combination for Guiding Peripheral Nerve Blocks: A Retrospective Registry Analysis. Anesth Analg. 2018 Oct;127(4):1035-1043. doi: 10.1213/ANE.0000000000003480. PMID 29863605
- [Background] Fredrickson MJ, Kilfoyle DH. Neurological complication analysis of 1000 ultrasound guided peripheral nerve blocks for elective orthopaedic surgery: a prospective study. Anaesthesia. 2009 Aug;64(8):836-44. doi: 10.1111/j.1365-2044.2009.05938.x. PMID 19604186
- [Derived] Oliver-Fornies P, Ortega Lahuerta JP, Gomez Gomez R, Gonzalo Pellicer I, Herranz Andres P, Sancho-Saldana A. Postoperative neurological complications after brachial plexus block: a retrospective study conducted at a teaching hospital. J Anesth. 2021 Dec;35(6):844-853. doi: 10.1007/s00540-021-02989-7. Epub 2021 Aug 25. PMID 34432155

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04451642/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04451642/ICF_001.pdf